CLINICAL TRIAL: NCT00710944
Title: An Open, Prospective, Controlled Study in the Maxilla to Evaluate Clinical Outcome of ASTRA TECH Implant System, OsseoSpeed™ Implants in Single Tooth Replacement Using an Immediate Loading Protocol in Extraction Sockets and Healed Ridges.
Brief Title: Study to Compare Survival for ASTRA TECH Implant System, OsseoSpeed™ Implants Following Immediate Loading in Extraction Sockets Versus Immediate Loading in Healed Ridges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-OSS-0006
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-06

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Jaw, Edentulous, Partially (missing/extracted/avulsed teeth in the maxilla within zone 15(4)-25(13))
MeSH Terms: conditions — Jaw, Edentulous, Partially; Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Extraction Sockets (Experimental): Immediate loading in extraction sockets.
  Interventions: Device: ASTRA TECH Implant System, OsseoSpeed™
- Healed Ridges (Experimental): Immediate loading in healed ridges.
  Interventions: Device: ASTRA TECH Implant System, OsseoSpeed™
- Grafted Sites (Experimental): Immediate loading of implants placed in grafted sites (four months healing after grafting).
  Interventions: Device: ASTRA TECH Implant System, OsseoSpeed™

INTERVENTIONS:
Device: ASTRA TECH Implant System, OsseoSpeed™ — ASTRA TECH Implant System, OsseoSpeed™: Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm.

SUMMARY:
The purpose of this study is to evaluate survival for ASTRA TECH Implant System, OsseoSpeed™ implants following immediate loading in extraction sockets versus immediate loading in healed ridges. Patients in need of single standing implants replacing teeth in the maxilla within zone 15-25 will be included and followed for 5 years. Primary objective is implant survival rate at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* 18 years of age and over
* A minimum of 20 stable intra occlusal contacts after planned restoration
* In need of single standing implants replacing missing / extracted / avulsed teeth in the maxilla within zone 15 to 25

Exclusion Criteria:

* Untreated rampant caries and uncontrolled periodontal disease
* Use of smoking tobacco at time of inclusion
* History of pre-surgical bone augmentation, within 4 months, in the planned implant area
* History of extraction without augmentation, within 3 months in the planned implant area
* Absence of opposing dentition
* Absence of adjacent (mesial and/or distal) natural tooth
* Uncontrolled diabetes
* Known pregnancy at time of inclusion
* Present alcohol or drug abuse
* Any systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Need for systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* Unable or unwilling to return for follow-up visits for a period of 5 years
* Unrealistic esthetical demands
* Unlikely to be able to comply with study procedures according to Investigators judgment
* Already included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Cooper, Prof, DDS, PhD, Principal Investigator — School of Dentistry, Chapel Hill
Locations (4):
- School of Dentistry, Chapel Hill, North Carolina, United States
- Dental School Department Periodontology, Ghent, Belgium
- Department of Oromaxillofacial Surgery, Hospital of the Christian- Albrechts University at Kiel, Kiel, Germany
- Universitat Internacional de Catalunya, Department de Odontología, Barcelona, Spain

REFERENCES:
- [Result] Cooper LF, Raes F, Reside GJ, Garriga JS, Tarrida LG, Wiltfang J, Kern M, de Bruyn H. Comparison of radiographic and clinical outcomes following immediate provisionalization of single-tooth dental implants placed in healed alveolar ridges and extraction sockets. Int J Oral Maxillofac Implants. 2010 Nov-Dec;25(6):1222-32. PMID 21197501
- [Result] Raes F, Cooper LF, Tarrida LG, Vandromme H, De Bruyn H. A case-control study assessing oral-health-related quality of life after immediately loaded single implants in healed alveolar ridges or extraction sockets. Clin Oral Implants Res. 2012 May;23(5):602-8. doi: 10.1111/j.1600-0501.2011.02178.x. Epub 2011 Apr 19. PMID 21504481
- [Result] De Bruyn H, Raes F, Cooper LF, Reside G, Garriga JS, Tarrida LG, Wiltfang J, Kern M. Three-years clinical outcome of immediate provisionalization of single Osseospeed() implants in extraction sockets and healed ridges. Clin Oral Implants Res. 2013 Feb;24(2):217-23. doi: 10.1111/j.1600-0501.2012.02449.x. Epub 2012 Apr 2. PMID 22469026
- [Result] Cooper LF, Reside GJ, Raes F, Garriga JS, Tarrida LG, Wiltfang J, Kern M, De Bruyn H. Immediate provisionalization of dental implants placed in healed alveolar ridges and extraction sockets: a 5-year prospective evaluation. Int J Oral Maxillofac Implants. 2014 May-Jun;29(3):709-17. doi: 10.11607/jomi.3617. PMID 24818212

RESULTS

PARTICIPANT FLOW:
Groups:
- Extraction Sockets: Immediate loading of implants placed in extraction sockets. OsseoSpeed™: OsseoSpeed™ Microthread™ Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm.
- Healed Ridges: Immediate loading of implants placed in healed ridges. OsseoSpeed™: OsseoSpeed™ Microthread™ Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm.
- Grafted Sites: Immediate loading of implants placed in grafted sites (four months healing after grafting).
  OsseoSpeed™: OsseoSpeed™ Microthread™ Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm.
Period: Overall Study
Arm/Group | Extraction Sockets | Healed Ridges | Grafted Sites
Started | 55 | 58 | 19
Completed | 45 | 49 | 17
Not Completed | 10 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Extraction Sockets: Immediate loading of implants placed in extraction sockets.
  ASTRA TECH Implant System, OsseoSpeed™: Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm.
- Healed Ridges: Immediate loading of implants placed in healed ridges.
  ASTRA TECH Implant System, OsseoSpeed™: Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm.
- Grafted Sites: Immediate loading of implants placed in grafted sites (four months healing after grafting).
  ASTRA TECH Implant System, OsseoSpeed™: Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm.
- Total: Total of all reporting groups
Arm/Group | Extraction Sockets | Healed Ridges | Grafted Sites | Total
Number analyzed (Participants) | 55 | 58 | 19 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (14) | 42 (15) | 40 (17) | 42 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 7 | 73
  Male | 22 | 25 | 12 | 59

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival
Description: An implant that has failed to osseointegrate, lost its osseointegration or fractured was considered a failure effective from the date of removal. The survival rate for individual implants was analyzed at each visit. Cumulative implant survival rate was calculated using Kaplan-Meier life-table estimation and reported as percentage of survived implants.
Time Frame: 12 months after implant placement
Population: Per protocol analysis presented, this includes implants immediately loaded (Group A: 55 implants in 55 subjects, Group B: 58 implants in 58 subjects, Group C: 19 implants in 19 subjects), of these 5 implants in total failed within 12 months after implant placement.
Measure: Number; unit: percentage of implants
Units Other Than Participants: Implants
Arm/Group | Extraction Sockets | Healed Ridges | Grafted Sites
Number analyzed (Participants) | 55 | 58 | 19
Number analyzed (Implants) | 55 | 58 | 19
percentage of implants | 94.55 | 98.28 | 94.73

ADVERSE EVENTS:
Groups:
- Extractions Sockets: Immediate loading of implants placed in extraction sockets. OsseoSpeed™: OsseoSpeed™ Microthread™ Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm.
Arm/Group | Extractions Sockets | Healed Ridges | Grafted Sites
Serious Adverse Events (participants affected / at risk) | 2/55 | 2/58 | 0/19
Other Adverse Events (participants affected / at risk) | 0/55 | 0/58 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Extractions Sockets (N=55) | Healed Ridges (N=58) | Grafted Sites (N=19)
Acute lymphangitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Prostate cancer (Reproductive system and breast disorders) | 1 | 0 | 0
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Stomach cancer (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less